CLINICAL TRIAL: NCT02884713
Title: Efficacy of Levofloxacin-Doxycycline Based Rescue Therapy for Helicobacter Pylori Eradication: A Prospective Open-label Trial in Saudi Arabia
Brief Title: Levofloxacin-Doxycycline for Helicobacter Pylori Eradication in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Fahad Alsohaibani, Consultant, Hepatology/Gastroenterology, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC # 2131064
Record Dates: First submitted 2016-08-11; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: GASTRITIS
MeSH Terms: conditions — Gastritis | interventions — Levofloxacin; Doxycycline; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levofloxacin and Doxycycline and Esomeprazole (Experimental): The rescue treatment was given for ten days consisting of levofloxacin 500 mg once daily, doxycycline 100 mg twice daily, and esomeprazole 20 mg twice daily
  Interventions: Drug: Levofloxacin; Drug: Doxycycline; Drug: Esomeprazole

INTERVENTIONS:
Drug: Levofloxacin — The primary objective was to evaluate the efficacy of the 10-day course of levofloxacin, doxycycline and esomeprazole in non-responders to first-line therapies for H. pylori eradication in Saudi Arabia. Secondary objectives included; symptoms response to treatment, factors associated with eradication of H. pylori and adverse events associated with the treatment
Drug: Doxycycline — The primary objective was to evaluate the efficacy of the 10-day course of levofloxacin, doxycycline and esomeprazole in non-responders to first-line therapies for H. pylori eradication in Saudi Arabia. Secondary objectives included; symptoms response to treatment, factors associated with eradication of H. pylori and adverse events associated with the treatment
Drug: Esomeprazole — The primary objective was to evaluate the efficacy of the 10-day course of levofloxacin, doxycycline and esomeprazole in non-responders to first-line therapies for H. pylori eradication in Saudi Arabia. Secondary objectives included; symptoms response to treatment, factors associated with eradication of H. pylori and adverse events associated with the treatment

SUMMARY:
Helicobacter pylori (H. pylori) eradication is achieved in 60-80% with first-line therapy. Different second-line therapeutic options are available. However, the success of second-line therapy has not been addressed or reported from Saudi Arabia.

Objectives The primary objective was to evaluate the efficacy of the 10-day course of levofloxacin, doxycycline and esomeprazole in non-responders to first-line therapies for H. pylori eradication in Saudi Arabia. Secondary objectives included; symptoms response to treatment, factors associated with eradication of H. pylori and adverse events associated with the treatment.

DETAILED DESCRIPTION:
A prospective, open-label, single arm study was conducted. Patients were recruited from a tertiary care hospital in Saudi Arabia from June 2013 to April 2014. A total of 55 patients had previously received standard triple therapy and/or sequential therapy in the period from 2011 to 2014 and failed to eradicate the infection. The rescue treatment was given for ten days consisting of levofloxacin 500 mg once daily, doxycycline 100 mg twice daily, and esomeprazole 20 mg twice daily. Urea-breath-test (UBT) was done at a minimum of 6 weeks after completion of the treatment to confirm the H. pylori eradication. Compliance and tolerability of the regimen were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Received previous treatment with triple therapy, sequential therapy or both
* Has evidence of persistence H. pylori infection by a positive urea breath test (UBT), histology or rapid urease test (HP Fast. GI supply™, PA, USA)

Exclusion Criteria:

* Previously treated with quadruple or levofloxacin-based therapy
* Had an allergy to doxycycline, levofloxacin or esomeprazole
* Pregnant or lactating
* Significant hepatic, renal, or cardiopulmonary disorders, or active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Eradication rate of second line levofloxacin- doxycycline based therapy for H. pylori eradication after failed fisrt line therapy using Urea Breath Test and its association with symptoms resolution. | 6 weeks
  The primary endpoint was a negative UBT after a minimum of 6 weeks after completion of treatment

SECONDARY OUTCOMES:
Symptoms response to treatment | 6 weeks
  Will use a visual analogue scale (VAS) on a questionnaire to look at the symptoms pre and post treatment and see if the eradication of h.pylori helped to resolve the symptoms
Factors associated with eradication of H.pylori | 6 weeks
  Physiological parameter: such as age and gender and prior use of triple or sequential therapy
Adverse events associated with the treatment | 6 weeks
  Will use a visual analogue scale (VAS) on a questionnaire (such as abdominal pain, headache, dizziness, and rash)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.